CLINICAL TRIAL: NCT03600701
Title: A Phase 2 Study of Atezolizumab and Cobimetinib in PD-1/PD-L1 Inhibitor Resistant or Refractory Non-Small Cell Lung Cancer
Brief Title: Atezolizumab and Cobimetinib in Treating Patients With Metastatic, Recurrent, or Refractory Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01812; NCI-2017-01812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10166 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10166 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2018-07-25; First posted 2018-07-26 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Refractory Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Biopsy; Specimen Handling; cobimetinib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (atezolizumab, cobimetinib) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on days 1, and cobimetinib PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Patients also undergo a CT scan, MRI, biopsy, and collection of blood throughout the trial.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cobimetinib; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC 0973; GDC-0973; GDC0973; MEK Inhibitor GDC-0973; XL 518; XL-518; XL518
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II trial studies how well atezolizumab and cobimetinib work in treating patients with non-small cell lung cancer that has spread from where it first started (primary site) to other places in the body (metastatic), has come back (recurrent), or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cobimetinib is used in patients whose cancer has a mutated (changed) form of a gene called BRAF. It is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps slow or stop the spread of cancer cells. Giving atezolizumab and cobimetinib may work better in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate durable overall response rate with atezolizumab plus cobimetinib in patients with metastatic non-small cell lung cancer (NSCLC) resistant or refractory to prior PD-1 or PD-L1 therapy.

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate of atezolizumab plus cobimetinib in patients with metastatic NSCLC resistant or refractory to prior PD-1 or PD-L1 therapy.

II. To evaluate the progression-free survival (PFS) of atezolizumab plus cobimetinib in patients with metastatic NSCLC resistant or refractory to prior PD-1 or PD-L1 therapy.

III. To evaluate the overall survival (OS) of atezolizumab plus cobimetinib in patients with metastatic NSCLC resistant or refractory to prior PD-1 or PD-L1 therapy.

IV. To evaluate the duration of response (DOR) of atezolizumab plus cobimetinib in patients with metastatic NSCLC resistant or refractory to prior PD-1 or PD-L1 therapy.

V. To evaluate the grade 3 and 4 toxicity rate in patients with metastatic NSCLC resistant or refractory to prior PD-1 or PD-L1 therapy when treated with atezolizumab plus cobimetinib.

EXPLORATORY OBJECTIVES:

I. To evaluate the consequences of treatment with atezolizumab plus cobimetinib on the tumor microenvironment in patients with metastatic NSCLC resistant or refractory to prior PD-1 or PD-L1 therapy.

II. To correlate genomic characteristics including tumor mutation burden to response to therapy with atezolizumab plus cobimetinib in patients with metastatic NSCLC resistant or refractory to prior PD-1 or PD-L1 therapy.

OUTLINE:

Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1 and cobimetinib orally (PO) once daily (QD) on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity. Patients also undergo a computed tomography (CT) scan, magnetic resonance imaging (MRI), biopsy, and collection of blood throughout the trial.

After completion of study treatment, patients are followed up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or recurrent non-small cell lung cancer (any histology is permitted)

  * Presence of a mutation in KRAS as detected by a Clinical Laboratory Improvement Act (CLIA)-approved assay is required for patients enrolled in cohort 1; central validation is not required for enrollment
  * Absence of a mutation in KRAS (KRAS wild type) is required for patients enrolled in cohort 2; central validation is not required for enrollment but KRAS mutation status must be known, regardless of histology
* Patients must have primary resistance to anti-PD-1 or anti-PD-L1 therapy, given as monotherapy or in combination with other agents; patients must have experienced progressive disease within 6 months (180 days) of initiating treatment with a PD-1/PD-L1 inhibitor

  * Anti-PD-1 or anti-PD-L1 therapy does not need to be the most recent therapy prior to study enrollment
* Patients with a sensitizing alteration in EGFR, ALK or ROS1 are eligible provided they have experienced disease progression or intolerance to treatment with an approved EGFR, ALK or ROS1 inhibitor, respectively; patients who have received investigational inhibitors may be eligible following discussion with the study principal investigator (PI)
* Patients must have disease amenable to core biopsy and be willing to undergo the required research biopsies
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam
* Age >= 18 years

  * Because no dosing or adverse event data are currently available on the use of atezolizumab in combination with cobimetinib in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 2,500/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x upper limit of normal [ULN] may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN (AST and/or ALT =< 5 x ULN for patients with liver involvement)
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN for patients with documented liver involvement or bone metastases)
* Creatinine clearance >= 30 mL/min/1.73 m^2 by Cockcroft-Gault
* Institutional normalized ratio (INR) and partial thromboplastin time (aPTT) =< 1.5 x ULN; (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose)
* Administration of atezolizumab or cobimetinib may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of study agent; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial

Exclusion Criteria:

* Patients who have not recovered from clinically significant adverse events (other than alopecia) due to prior anti-cancer therapy
* Treatment with any investigational agent within 4 weeks prior to cycle 1, day 1
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients with symptomatic central nervous system (CNS) metastases are excluded

  * Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met:

    * Evaluable or measurable disease outside the CNS
    * No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
    * No history of intracranial hemorrhage or spinal cord hemorrhage
    * No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted
    * No neurosurgical resection or brain biopsy within 28 days prior to cycle 1, day 1
  * Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

    * Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
    * No stereotactic radiation or whole-brain radiation within 28 days prior to cycle 1, day 1
    * Screening CNS radiographic study >= 4 weeks from completion of radiotherapy and >= 2 weeks from discontinuation of corticosteroids
* Has a known concurrent malignancy that is expected to require active treatment within two years, or may interfere with the interpretation of the efficacy and safety outcomes of this study in the opinion of the treating investigator; superficial bladder cancer, non-melanoma skin cancers, or low grade prostate cancer not requiring therapy should not exclude participation in this trial
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to atezolizumab or cobimetinib
* History of congenital long QT syndrome or corrected QT interval (QTc) by Fridericia Formula > 450 msec within 28 days of cycle 1, day 1
* Cardiac ejection fraction below institutional lower limit of normal (LLN) or below 50%, whichever is lower, as determined by echocardiogram or multigated acquisition (MUGA) scan within 4 weeks of cycle 1, day 1
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, central serous chorioretinopathy, retinal vein occlusion (RVO), or neovascular macular degeneration
* Any grade 3 or above hemorrhage or bleeding event within 4 weeks prior to initiation of study treatment
* History of stroke, reversible ischemic neurological defect, or transient ischemic attack within 6 months prior to initiation of study treatment
* Patients receiving any medications or substances that are strong or moderate inhibitors or inducers of CYP3A4 enzymes are ineligible; these include St. John's wort or hyperforin (potent CYP3A4 enzyme inducer) and grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor); because the lists of these agents are constantly changing, it is important to regularly consult medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, autoimmune hemolytic anemia, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Any significant active infection requiring treatment within 14 days prior to cycle 1, day 1
* Major surgical procedure within 28 days prior to cycle 1, day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study
* Uncontrolled pleural or pericardial effusion or ascites requiring recurrent drainage procedures
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active tuberculosis (TB), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because both atezolizumab and cobimetinib are expected to cause fetal harm if used during pregnancy; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cobimetinib or atezolizumab, breastfeeding should be discontinued if the mother is treated with either therapy; these potential risks may also apply to other agents used in this study
* Inability or unwillingness to swallow pills
* History of malabsorption syndrome or other condition that would interfere with enteral absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2026-10-03 (Estimated)

PRIMARY OUTCOMES:
Durable response rate to therapy | Up to 90 days
  Will be presented with descriptive statistics. A durable response is defined as a response meeting Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria in a patient whose response duration was of at least 6 months.

SECONDARY OUTCOMES:
Overall response rate | Up to 90 days
  Will be assessed using RECIST version 1.1 criteria. Will use chi-square statistics to describe and analyze results with ethnic categories and racial categories, respectively.
Duration of response | Up to 90 days
Progression free survival (PFS) | Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 90 days
  Kaplan-Meier estimates will be used to describe the PFS. The association of PFS with biomarkers will be assessed using Cox regression model with model adequacy assessment.
Overall survival (OS) | From start of study treatment to time of death, assessed up to 90 days
  Kaplan-Meier estimates will be used to describe the OS. The association of survival with biomarkers will be assessed using Cox regression model with model adequacy assessment.
Grade 3 and 4 toxicities | Up to 90 days
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.
Biomarker analysis | Up to 90 days
  The analysis of biomarkers will also be descriptive given the limited sample sizes. Categorical data analysis methods such as Chi-square will be used to evaluate the correlation of baseline tumor mutation burden to response to therapy. Regression and correlation will be used for assessing the association between continuous variables such as tumor burden and other markers and patient characteristics such as age.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen V Liu, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (18):
- United States (18):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UC San Diego Moores Cancer Center, La Jolla, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYP/Weill Cornell Medical Center, New York, New York
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Hayworth Cancer Center, High Point, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia